CLINICAL TRIAL: NCT00396279
Title: An Open-Label, Multi-Center, Phase 2 Safety and Efficacy Study of Denosumab (AMG 162) in Subjects With Recurrent or Unresectable Giant Cell Tumor (GCT) of Bone
Brief Title: Safety and Efficacy Study of Denosumab in Patients With Recurrent or Unresectable Giant Cell Tumor of Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040215
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: GCT; Giant Cell Tumor of Bone
Keywords: Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab; Calcium; Vitamin D

ARMS (1):
- Denosumab (Experimental): Participants received denosumab 120 mg once every 4 weeks (Q4W), with an additional 120 mg doses on Days 8 and 15 of the first month of treatment. All participants were instructed to take daily supplements of at least 500 mg of calcium and 400 IU of vitamin D. Participants were to continue to receive denosumab until one of the following occurred: complete tumor resection, disease progression without clinical benefit, or decision by the participant to discontinue for any reason.
  Interventions: Biological: Denosumab; Dietary Supplement: Calcium/Vitamin D

INTERVENTIONS:
Biological: Denosumab — Administered by subcutaneous injection
  Other Names: Xgeva®
Dietary Supplement: Calcium/Vitamin D

SUMMARY:
To determine how safe and effective denosumab is in treating patients with giant cell tumor of bone.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years and older
* Histologically confirmed and measurable giant cell tumor (GCT)
* Recurrent GCT confirmed by radiology or unresectable GCT
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Pateints for whom surgery to the affected limb/area is planned within 27 days after receiving 1st dose of denosumab
* Radiation to affected region within 28 days before enrollment to study
* Known diagnosis of osteosarcoma or brown tumor of bone
* Known history of second malignancy within the past 5 years, except for basal cell carcinoma or cervical carcinoma in situ
* Concurrent treatment with bisphosphonates, calcitonin, or interferon.

Other criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-07-10 (Actual); Primary Completion 2008-04-07 (Actual); Study Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Branstetter DG, Nelson SD, Manivel JC, Blay JY, Chawla S, Thomas DM, Jun S, Jacobs I. Denosumab induces tumor reduction and bone formation in patients with giant-cell tumor of bone. Clin Cancer Res. 2012 Aug 15;18(16):4415-24. doi: 10.1158/1078-0432.CCR-12-0578. Epub 2012 Jun 18. PMID 22711702
- [Background] Thomas D, Henshaw R, Skubitz K, Chawla S, Staddon A, Blay JY, Roudier M, Smith J, Ye Z, Sohn W, Dansey R, Jun S. Denosumab in patients with giant-cell tumour of bone: an open-label, phase 2 study. Lancet Oncol. 2010 Mar;11(3):275-80. doi: 10.1016/S1470-2045(10)70010-3. Epub 2010 Feb 10. PMID 20149736
- [Derived] Engellau J, Seeger L, Grimer R, Henshaw R, Gelderblom H, Choy E, Chawla S, Reichardt P, O'Neal M, Feng A, Jacobs I, Roberts ZJ, Braun A, Bach BA. Assessment of denosumab treatment effects and imaging response in patients with giant cell tumor of bone. World J Surg Oncol. 2018 Sep 19;16(1):191. doi: 10.1186/s12957-018-1478-3. PMID 30231890
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 10 July 2006; Last patient enrolled 25 January 2008. Results data are reported as of the data cut-off date of 07 April 2008.
Groups:
- Denosumab: Participants received denosumab 120 mg once every 4 weeks (Q4W), with an additional 120 mg dose on Days 8 and 15 of the first month of treatment. All participants were instructed to take daily supplements of at least 500 mg of calcium and 400 IU of vitamin D. Participants were to continue to receive denosumab until one of the following occurred: complete tumor resection, disease progression without clinical benefit, or decision by the participant to discontinue for any reason.
Period: Overall Study
Arm/Group | Denosumab
Started | 37
Completed | 7 (Defined as participants with a complete resection)
Not Completed | 30
Not completed — Ongoing in study | 26
Not completed — Disease progression | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Denosumab
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 27
  Black or African American | 2
  Hispanic or Latino | 5
  Asian | 3
Giant Cell Tumor Disease Type [Number; unit: participants]
  Primary unresectable | 13
  Recurrent unresectable | 18
  Recurrent resectable | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — 0: Fully active, able to carry on all pre-disease performance without restriction;
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work;
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours;
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours;
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  participants
    0 - Fully Active | 13
    1 - Restricted but ambulatory | 21
    2 - Ambulatory but unable to work | 1
    3 - Limited selfcare, confined to bed >50% daytime | 0
    4 - Completely disabled | 0
    Missing | 2
Percent of giant cells in tumor on pre-treatment biopsy [Mean (Standard Deviation); unit: percentage of giant cells in tumor] | 28.7 (16.1)
Location of target lesion [Number; unit: participants]
  Lower extremities | 8
  Upper extremities | 5
  Pelvis | 9
  Spine | 3
  Pulmonary disease | 9
  Dorsal vertebrae | 1
  Pelvic region | 1
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Giant Cell Tumor Response
Description: A treatment response was defined for participants with tissue samples obtained and measured by histopathology as: • at least 90% elimination of giant cells relative to Baseline, or • complete elimination of giant cells in cases where giant cells represent < 5% of tumor cells. A response was defined for participants who have only radiographs (histopathology not available) as lack of progression of the target lesion at week 25 by radiographic measurements compared with Baseline. For participants with both a core biopsy and resected tissue obtained, the sample closest to week 25 was used in the analysis.
Time Frame: From enrollment until 25 weeks
Population: The efficacy analysis set included participants with a Baseline histology assessment and at least 1 postdose histology assessment from weeks 5-25; or a Baseline radiology assessment and at least 1 postdose radiology assessment from weeks 5-25. Evaluable participants had to be on study for at least 28 days after administration of the first dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Denosumab
Number analyzed (Participants) | 35
percentage of participants | 85.7 [69.7 to 95.2]

2. Secondary Outcome: Percent Change From Baseline in Urinary N-telopeptide Corrected for Urine Creatinine
Description: Urinary N-telopeptide (of type 1 collagen) corrected for urine creatinine (uNTX/Cr) is a bone turnover marker used to measure the activity of denosumab. Percent change from Baseline in uNTX/Cr was measured over time.
Time Frame: Baseline and Weeks 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, and 81
Population: Efficacy Analysis Set with available data at each time point (n).
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Denosumab
Number analyzed (Participants) | 35
percent change
  Week 5 (n=30) | -70.9 [-79.6 to -15.0]
  Week 9 (n=29) | -77.0 [-85.7 to -42.9]
  Week 13 (n=27) | -60.0 [-84.2 to -36.0]
  Week 17 (n=26) | -59.5 [-79.3 to -37.1]
  Week 21 (n=24) | -64.5 [-80.1 to -19.1]
  Week 25 (n=20) | -56.4 [-76.2 to 3.6]
  Week 29 (n=21) | -52.8 [-78.4 to -22.8]
  Week 33 (n=15) | -35.0 [-83.8 to 22.0]
  Week 37 (n=13) | -71.1 [-83.4 to -41.4]
  Week 41 (n=11) | -57.3 [-78.1 to -22.4]
  Week 45 (n=8) | -59.1 [-81.8 to -47.5]
  Week 49 (n=7) | -59.0 [-74.0 to -0.9]
  Week 53 (N=8) | -49.0 [-81.5 to -29.3]
  Week 57 (n=6) | -65.1 [-78.4 to -21.9]
  Week 61 (n=3) | -59.2 [-92.5 to 23.1]
  Week 65 (n=3) | -69.2 [-79.6 to 33.2]
  Week 69 (n=4) | -64.2 [-88.8 to -13.4]
  Week 73 (n=1) | -47.5 [-47.5 to -47.5]
  Week 77 (n=2) | -76.8 [-86.8 to -66.7]
  Week 81 (n=2) | -13.3 [-53.8 to 27.1]

3. Secondary Outcome: Percent Change From Baseline in Serum C-terminus Peptide (of Type 1 Collagen)
Description: Serum C-terminus peptide (of type 1 collagen; CTX1) is a bone turnover marker used to measure the activity of denosumab. Percent change from Baseline in CTX was measured over time.
Time Frame: Baseline and Weeks 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 53, 57, 61, 65, 69, 73, 77, and 81
Population: Efficacy Analysis Set with available data at each time point (n).
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Denosumab
Number analyzed (Participants) | 35
percent change
  Week 5 (n=33) | -78.9 [-85.2 to -71.2]
  Week 9 (n=33) | -79.8 [-87.9 to -66.1]
  Week 13 (n=31) | -80.4 [-85.7 to -71.3]
  Week 17 (n=28) | -82.6 [-85.2 to -70.4]
  Week 21 (n=26) | -82.0 [-87.0 to -66.4]
  Week 25 (n=24) | -79.5 [-86.5 to -69.2]
  Week 29 (n=21) | -82.8 [-85.2 to -60.3]
  Week 33 (n=16) | -74.8 [-83.2 to -59.0]
  Week 37 (n=14) | -82.4 [-87.0 to -69.6]
  Week 41 (n=10) | -86.1 [-89.6 to -58.5]
  Week 45 (n=8) | -79.6 [-86.4 to -70.0]
  Week 49 (n=7) | -82.0 [-90.0 to -76.7]
  Week 53 (N=8) | -87.3 [-89.8 to -84.2]
  Week 57 (n=6) | -86.2 [-87.7 to -85.2]
  Week 61 (n=4) | -84.9 [-88.3 to -83.0]
  Week 65 (n=3) | -83.5 [-87.0 to -77.5]
  Week 69 (n=4) | -84.2 [-86.9 to -80.0]
  Week 73 (n=2) | -81.9 [-85.2 to -78.5]
  Week 77 (n=2) | -84.2 [-87.5 to -80.9]
  Week 81 (n=2) | -84.9 [-89.6 to -80.3]

4. Secondary Outcome: Serum Denosumab Trough Concentrations
Description: Serum concentrations of denosumab were measured by a validated conventional sandwich enzyme-linked immunosorbent assay (ELISA).
Time Frame: Blood samples were collected on Days 1 (baseline), 8, 15 and Weeks 5 (Day 29), 9, 13, 25, and 49.
Population: The pharmacokinetics analysis set included participants who received at least 1 dose of denosumab and for whom at least 1 serum denosumab trough concentration was available. 'n' indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab
Number analyzed (Participants) | 37
ng/mL
  Day 1 (n=32) | NA (NA) — Below the lower limit of quantification
  Day 8 (n=32) | 19000 (24100)
  Day 15 (n=28) | 31600 (27300)
  Day 29 (n=33) | 36400 (20600)
  Week 9 (n=32) | 27500 (17300)
  Week 13 (n=25) | 23300 (12400)
  Week 25 (n=23) | 19900 (9700)
  Week 49 (n=9) | 21400 (8900)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is defined as an undesirable medical occurrence (e.g., sign, symptom, or diagnosis) or worsening of a pre-existing medical condition. A serious adverse event (SAE) is defined by regulatory authorities as one that • is fatal • is life threatening (places the participant at immediate risk of death) • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect • other significant medical hazard. The severity of adverse events was assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, version 3.0) based on the following general guideline: Grade 1: Mild AE Grade 2: Moderate AE Grade 3: Severe AE Grade 4: Life-threatening or disabling AE Grade 5: Death related to AE. AEs were assessed by the Investigator for relatedness to study drug.
Time Frame: From the first dose of study drug until the data cut-off date of April 7 2008; a maximum of 18 months
Population: All participants who received at least 1 dose of denosumab.
Measure: Number; unit: participants
Arm/Group | Denosumab
Number analyzed (Participants) | 37
participants
  Any AE | 33
  Serious AE | 5
  Fatal AE | 1
  AE leading to study discontinuation | 2
  AE leading to study drug discontinuation | 3
  CTCAE Grade 3, 4, or 5 | 5
  Any AE related to study drug | 10

6. Secondary Outcome: Number of Participants With Anti-Denosumab Antibodies
Description: Validated immunoassays were used to test for the presence of anti-denosumab antibodies throughout the study.
Time Frame: From enrollment until the data cut-off date of April 7 2008; a maximum time of 18 months.
Population: Participants who received at least 1 dose of denosumab and had at least 1 anti-denosumab antibody sample.
Measure: Number; unit: participants
Arm/Group | Denosumab
Number analyzed (Participants) | 31
participants | 0

ADVERSE EVENTS:
Time Frame: up to 1 year 6 months
Description: The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency.
Groups:
- Denosumab 120 mg Q4W: Participants received a dose loading regimen of 3 subcutaneous injections of denosumab 120 mg every week for 3 weeks (study Days 1, 8, and 15), followed by a week of rest, and then 120 mg denosumab once every 4 weeks (Q4W) from Day 29.
Arm/Group | Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 5/37
Other Adverse Events (participants affected / at risk) | 25/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W (N=37)
Nausea (Gastrointestinal disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg Q4W (N=37)
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Fatigue (General disorders) | 3
Bronchitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.